CLINICAL TRIAL: NCT06142539
Title: The Impact of Different Scanning Methods and Reconstruction Algorithms on CT Image Quality
Status: Recruiting | Type: Observational
Sponsor: Wei Li (Other)
Responsible Party: Sponsor-Investigator, Wei Li, clinical professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: WLi
Record Dates: First submitted 2023-11-07; First posted 2023-11-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: CT Examination of the Abdomen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SDCT group
- LDCT group
  Interventions: Radiation: CT Radiation Doses

INTERVENTIONS:
Radiation: CT Radiation Doses — Obtaining Low CT Radiation Doses by Adjusting Dose Levels
  Groups: LDCT group

SUMMARY:
Purpose: To evaluate the image quality of deep learning-based image reconstruction (DLIR) algorithm in unenhanced abdominal low-dose CT (LDCT).

Methods: CT images of a phantom were reconstructed with Hybrid iterative reconstruction and deep learning image reconstruction (DLIR). The noise power spectrum (NPS) and task transfer function (TTF) were measured. Two patient groups were included in this study: consecutive patients who underwent unenhanced abdominal standard-dose CT reconstructed with hybrid iterative reconstruction (SDCT group) and consecutive patients who underwent unenhanced abdominal LDCT reconstructed of HIR and DLIR (LDCT group). The CT values, standard deviation (SD), signal-to-noise ratio (SNR), and contrast-to-noise ratio (CNR) of the hepatic parenchyma and paraspinal muscle and abdominal subcutaneous fat were evaluated. Radiologists assessed the subjective image quality and lesion diagnostic confidence using a 5-point Likert scale. Quantitative and qualitative parameters were compared between SDCT and LDCT groups.

ELIGIBILITY:
Inclusion Criteria:

Abdominal CT examination

Exclusion Criteria:

pregnancy and lactation for women unstable breath holding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Abdominal CT examination
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Results of phantom research | up to six months
  Compare the changes in spatial resolution (TTF curve) and noise (NPS curve) between different algorithms
Results of human clinical study | up to six months
  General information of clinical trial personnel Compare the general information of two groups of subjects, such as age, weight（kg）, height（m）, gender, and BMI (kg/m2).
  Quantitative image analysis The standard deviation (SD), signal-to-noise ratio (SNR), and contrast-to-noise ratio (CNR) of the hepatic parenchyma and paraspinal muscle were evaluated.
  Qualitative image analysis Two radiologists qualitatively assessed the overall image noise and overall image quality depiction.

SECONDARY OUTCOMES:
Patient demographics | up to six months
  Participant demographics: Age (year)/Gender/Body weight (kg) / Body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- uCT960+, Shandong, Jinan Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi H, Cui D, Xu S, Li W, Zeng Q. Image quality assessment of artificial intelligence iterative reconstruction for low dose unenhanced abdomen: comparison with hybrid iterative reconstruction. Abdom Radiol (NY). 2025 Jul;50(7):3353-3362. doi: 10.1007/s00261-024-04760-4. Epub 2024 Dec 21. PMID 39707032